CLINICAL TRIAL: NCT02252510
Title: Evaluation of the Reliability for the Measurement of Sperm DNA Damage by a Sperm Chromatin Dispersion Test (Halosperm)
Brief Title: Reliability for the Detection of Sperm DNA Damage by a Sperm Chromatin Dispersion Test (Halosperm)
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0208
Record Dates: First submitted 2014-09-26; First posted 2014-09-30 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Infertile Men

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Other: HALOSPERM

SUMMARY:
It is proposed to measure sperm DNA damage by sperm chromatin dispersion test. This measurement helps to better diagnose male infertility and seems easy to apply in routine. However, the reliability of this method needs to be evaluated before applying for clinical practice in andrology laboratory.

DETAILED DESCRIPTION:
The aim of this study is to measure the inter and intra-observer reliability for the measurements of sperm DNA damage by sperm chromatin dispersion test (halosperm). The gold standard to measure sperm DNA damage is TUNEL (Terminal desoxynucleotidyl end labelling) method. However, this method is not easy to apply in routine. Therefore we investigate to analyse the inter-method reliability between sperm chromatin dispersion test and TUNEL.

ELIGIBILITY:
Inclusion Criteria:

* infertile men
* <50 years
* with at least 5.106spermatozoa/ml in the ejacu

Exclusion Criteria:

* azoospermia

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: infertile men
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
- Percentage of spermatozoa with DNA damage (Sperm chromatin dispersion test) | at day 1

SECONDARY OUTCOMES:
Percentage of sperm DNA damage measured by TUNEL method | at day 1